CLINICAL TRIAL: NCT00689611
Title: Zyban as an Effective Smoking Cessation Aid for Patients Following an Acute Coronary Syndrome: The ZESCA Trial
Acronym: ZESCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mark Eisenberg (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor-Investigator, Mark Eisenberg, MD, MPH, Professor of Medicine, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZESCA 9197; ISRCTN75356261
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Smoking
Keywords: Acute coronary syndrome; Myocardial infarction; Smoking cessation; Zyban; Secondary intervention post-ACS
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Smoking; Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P (Placebo Comparator): Half of patients will receive placebo for 9 weeks.
  Interventions: Drug: Placebo
- A (Active Comparator): Half of patients will receive bupropion for 9 weeks.
  Interventions: Drug: Bupropion HCl ER

INTERVENTIONS:
Drug: Bupropion HCl ER — 150 mg tablets po qd for 3 days and then 150 mg po bid for remainder of 9 weeks
  Other Names: Zyban
  Arms: A
Drug: Placebo — Placebo
  Arms: P

SUMMARY:
Patients who continue to smoke after a heart attack have a 35% increased risk of a recurrent event or death compared with those who quit. Many patients attempt to stop smoking after a heart attack, but relapse rates approach 66%. A variety of smoking cessation aids have been shown to be effective for the general population. However, bupropion is the only non-nicotine replacement therapy shown to improve abstinence rates in healthy young smokers. Furthermore, nicotine replacement therapies (NRTs) are contraindicated in the immediate period following a heart attack because of the undesirable effects of nicotine. Although bupropion has been successfully used to reduce smoking rates in healthy young populations, its efficacy and safety in the setting of patients recovering from an ACS is unknown. These patients, if they continue to smoke, are at exceptionally high risk for recurrent cardiac events. If bupropion is effective in this population, it will have a major impact on secondary prevention of recurrent clinical events in patients who suffer a heart attack.

DETAILED DESCRIPTION:
Patients who continue smoking after ACS have a 35% increased risk of reinfarction or death compared with those who quit. Many patients attempt to stop smoking after an acute coronary syndrome (ACS), but relapse rates approach 66%. A variety of smoking cessation aids have been shown to be effective for the general population. However, physicians are reluctant to use a nicotine-based therapy because of its hemodynamic effects. Bupropion is the only non-nicotine replacement therapy shown to improve abstinence rates in healthy young smokers by approximately 50%. Although bupropion has successfully been used to reduce smoking rates in healthy young populations, its efficacy and safety in the setting of patients recovering from an ACS is unknown.

The ZESCA Trial will directly compare the efficacy and safety of bupropion versus placebo as a means of reducing smoking rates in patients following an ACS. The ZESCA Trial will be a multi-center effort, coordinated from the Jewish General Hospital/McGill University (Montreal, Quebec). A total of 1500 patients will be randomized following an ACS but before hospital discharge via an Internet web site. Prior to the start of the treatment, patients in both treatment arms will receive a standard physician-administered counseling session regarding smoking cessation. Patients will begin treatment in-hospital and will be monitored in-hospital for ≥ 2 days prior to discharge. Half the patients will receive bupropion for 9 weeks and the other half will receive placebo pills for 9 weeks. Patients receiving bupropion will take 150 mg once per day for 3 days and then 150 mg twice per day for the remainder of 9 weeks. Prior to discharge, the patients will receive an information sheet listing the possible side effects of bupropion. They will be advised to consult the treating physician should they experience any listed side effects. While in-hospital, patients will have quit smoking and they will be instructed to not restart smoking when discharged. Phone calls to the patients will be made by the study nurses at weeks 1 and 2 of the 9-week treatment period. In addition, the patients will have clinic visits at weeks 4 and 9 as well as months 6 and 12. Smoking abstinence will be assessed at 4 weeks, 9 weeks, 6 months, and 12 months after randomization. Smoking abstinence will be defined as the complete abstinence in the week prior to the clinic visits and levels of exhaled carbon monoxide ≤ 10 ppm. Side effects of bupropion in patients following ACS as well as clinical events following initiation of treatment will be measured at weeks 1-8 (by telephone calls), and weeks 4 and 9 as well as months 6 and 12 (by clinic visits). Withdrawal symptoms will also be assessed by the nurses during their weekly calls.

Trials previously conducted with bupropion involved young healthy smokers. The ZESCA trial will be the first to examine the utility of bupropion in a group of patients with an ACS. These patients, if they continue to smoke, are at exceptionally high risk for recurrent cardiac events. If bupropion is effective in this population, it will have a major impact on secondary prevention of recurrent clinical events in patients who suffer an ACS.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Smoke at least 10 cigarettes/day for the past year
* Suffered an enzyme-positive ACS
* Planned hospitalization of ≥24 hours
* Motivated to quit smoking
* Likely to be available for follow-up
* Able to understand and read English or French

Exclusion Criteria:

* Medical condition with a prognosis of < 1 year
* Pregnant or lactating
* Current use of Wellbutrin or any other medications that contain bupropion
* Current use of any medical therapy for smoking cessation (e.g. BuSpar, fluoxetine, doxepin, nicotine gum, or nicotine patch)
* Current seizure disorder, history of seizures or predisposition to seizures (e.g. history of brain tumor, severe head trauma, or stroke)
* History of bulimia or anorexia nervosa
* Current diagnosis of major depression (requiring medication), bipolar disease, or dementia
* History of suicidal events (previous suicide attempt, suicidal ideation) or family history of suicide
* Diagnosed hepatic failure, cirrhosis, hepatitis or history of hepatic impairment (AST or ALT levels ≥ 2 times upper limit of normal prior to admission for ACS)
* Renal impairment with creatinine levels ≥ 2 times the upper limit of normal
* Excessive alcohol consumption defined as ≥ 14 alcoholic drinks per week
* Use of any illegal drugs in the past year (e.g. cocaine, heroin, opiates)
* Current use of medications that lower seizure threshold e.g. amantadine, anti-depressants, anti-malarials, anti-psychotics, levodopa, lithium, quinolone antibiotics, ritonavir, systemic steroids, theophyllin, type 1C antiarrhythmics (e.g. encainide, flecainide, propafenone)
* Use of MAO inhibitors or thioridazine in the past 15 days
* Current use of over-the-counter stimulants (e.g. ephedrine, phenylephrine) or anoretics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2005-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Eisenberg, MD, MPH, Principal Investigator — Jewish General Hospital/ McGill University
Locations (38):
- United States (13):
  - Parkview Medcial Center, Pueblo, Colorado
  - Central Maine Medical Center, Lewiston, Maine
  - Bay Regional Medical Center, Bay City, Michigan
  - Bassett Healthcare, Cooperstown, New York
  - United Health Services, Johnson City, New York
  - Stony Brook Hospital and Medical Center, Stony Brook, New York
  - Schuster Cardiology, Kettering, Ohio
  - Southwest Cardiology, Kettering, Ohio
  - DVA Medical Center, Oklahoma City, Oklahoma
  - Advanced Cardiology Specialists, Scranton, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Riverside Hospital, Newport News, Virginia
  - Charleston Area Medical Center, South Charleston, West Virginia
- National Heart Foundation of Bangladesh, Dhaka, Bangladesh
- Canada (20):
  - Peter Lougheed Centre of the Calgary General Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Victoria General Hospital, Winnipeg, Manitoba
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - New Brunswick Heart Centre, Saint Johns, New Brunswick
  - Valley Regional Hospital, Kentville, Nova Scotia
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hopital de la Cite de la Sante, Laval, Quebec
  - CHA Hotel-Dieu de Levis, Lévis, Quebec
  - SMBD- Jewish General Hospital, Montreal, Quebec
  - Hopital Sacre-Coeur de Montreal, Montreal, Quebec
  - Hotel-Dieu, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Hopital Laval, Québec, Quebec
  - Hopital Fleurimont, Sherbrooke, Quebec
  - CSSS de Sorel-Tracy, Sorel-Tracy, Quebec
  - CSSS de la Region de Thetford, Thetford-Mines, Quebec
  - Saskatchewan Drug Research Institute, Saskatoon, Saskatchewan
- Centre for Chronic Disease Control, New Delhi, India
- Isfahan Cardiovascular Research Centre, Isfahan, Iran, Iran
- InterActive Research and Development, Karachi, Pakistan
- University Hospital F. Bourguiba, Sousse, Sousse Governorate, Tunisia

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Taylor GM, Lindson N, Farley A, Leinberger-Jabari A, Sawyer K, Te Water Naude R, Theodoulou A, King N, Burke C, Aveyard P. Smoking cessation for improving mental health. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD013522. doi: 10.1002/14651858.CD013522.pub2. PMID 33687070
- [Derived] Zhang DD, Eisenberg MJ, Grandi SM, Joseph L, O'Loughlin J, Paradis G, Lozano P, Filion KB. Bupropion, smoking cessation, and health-related quality of life following an acute myocardial infarction. J Popul Ther Clin Pharmacol. 2014;21(3):e346-56. Epub 2014 Oct 8. PMID 25326910
- [Derived] Shimony A, Grandi SM, Pilote L, Joseph L, O'Loughlin J, Paradis G, Rinfret S, Sarrafzadegan N, Adamjee N, Yadav R, Gamra H, Diodati JG, Eisenberg MJ; ZESCA Investigators. Utilization of evidence-based therapy for acute coronary syndrome in high-income and low/middle-income countries. Am J Cardiol. 2014 Mar 1;113(5):793-7. doi: 10.1016/j.amjcard.2013.11.024. Epub 2013 Dec 12. PMID 24440324

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo for 9 weeks.
- Bupropion: Participants received bupropion for 9 weeks.
  Bupropion HCl ER: 150 mg tablets po qd for 3 days and then 150 mg po bid for remainder of 9 weeks.
Period: Overall Study
Arm/Group | Placebo | Bupropion
Started | 200 | 192
Completed | 159 | 146
Not Completed | 41 | 46
Not completed — Death | 6 | 9
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Lost to Follow-up | 27 | 28

BASELINE CHARACTERISTICS:
Population: All enrolled participants were included in the baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bupropion | Total
Number analyzed (Participants) | 200 | 192 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.3) | 54.5 (10.4) | 53.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 65
  Male | 166 | 161 | 327
Region of Enrollment [Number; unit: participants]
  United States | 35 | 33 | 68
  Pakistan | 18 | 18 | 36
  Canada | 101 | 96 | 197
  Iran, Islamic Republic of | 31 | 31 | 62
  Tunisia | 6 | 4 | 10
  India | 9 | 10 | 19
No. of years smoked [Mean (Standard Deviation); unit: years] | 32.6 (11.9) | 33.2 (13.0) | 32.9 (12.4)
No. of cigarettes/day (past year) [Mean (Standard Deviation); unit: cigarettes/day] | 23.2 (10.4) | 23.2 (10.8) | 23.2 (10.6)
Index admission was for ST-segment elevation myocardial infarction [STEMI] [Number; unit: participants] | 133 | 121 | 254
Cardiac catheterization during index admission [Number; unit: participants] | 136 | 128 | 264
Percutaneous coronary intervention during index admission [Number; unit: participants] | 104 | 93 | 197
Coronary artery bypass graft during index admission [Number; unit: participants] | 15 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: The primary end point was 7-day point prevalence smoking abstinence at 12 months. Smoking cessation was defined as self-reported abstinence in the week before the 12-month clinic visit and a measurement of exhaled carbon monoxide less than 11 ppm.
  The primary end point was analyzed on an intention-to-treat (ITT) basis. Our ITT analysis assumed that those who withdrew consent or were lost to follow-up had returned to smoking at their baseline rates. This assumption is common in smoking cessation trials.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bupropion
Number analyzed (Participants) | 194 | 183
percentage of participants | 32.0 | 37.2

2. Secondary Outcome: Composite Major Adverse Cardiovascular Events (MACE)
Description: All clinical end points were adjudicated by members of the Endpoints Evaluation Committee who were blinded to treatment assignment.
  Composite MACE (death, myocardial infarction, unstable angina)
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bupropion
Number analyzed (Participants) | 200 | 192
percentage of participants | 11.0 | 13.0

ADVERSE EVENTS:
Arm/Group | Placebo | Bupropion
Serious Adverse Events (participants affected / at risk) | 37/200 | 34/192
Other Adverse Events (participants affected / at risk) | 48/200 | 58/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=200) | Bupropion (N=192)
Death (General disorders) | 6 (6) | 9 (9) — Deaths due to: coronary dissection, cardiac arrest (2), multisystem organ failure post-CABG, complications related to duodenal perforation and recurrent septic shock, ischemic event in the bowel or spinal cord.
Myocardial Infarction (Cardiac disorders) | 5 (5) | 5 (5)
Unstable Angina (Cardiac disorders) | 11 (11) | 12 (12)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Psychiatric event (Psychiatric disorders) | 1 (1) | 2 (2) — Includes delirium, hallucination, and suicidal ideation
Other (General disorders) | 17 (17) | 9 (9) — Specific adverse event terms by treatment group are unknown.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=200) | Bupropion (N=192)
Insomnia (Nervous system disorders) | 36 (36) | 43 (43)
Dry mouth (General disorders) | 18 (18) | 26 (26)
Dizziness (General disorders) | 17 (17) | 15 (15)
Dysgeusia (General disorders) | 13 (13) | 16 (16)
Constipation (Gastrointestinal disorders) | 12 (12) | 14 (14)
Dream abnormality (General disorders) | 17 (17) | 7 (7)
Pruritus (General disorders) | 8 (8) | 5 (5)

LIMITATIONS AND CAVEATS:
Relatively high number who withdrew or were lost to follow-up (22.2%), but within expectations for smoking cessation trials; Relatively small numbers of serious adverse events occurred, limiting power to examine secondary safety end points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less